CLINICAL TRIAL: NCT02104297
Title: The Effect of Deksmedetomidin and Remifentanil Infusion on Extubation Agitation and Recovery Conditions on Nasal Septoplasty Operation
Brief Title: Effect of Deksmedetomidine and Remifentanil in Extubation Agitation
Acronym: EA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Medical Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Agitation
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Agitation
Keywords: Nasal septum operation; agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Dexmedetomidine; Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deksmedetomidine infusion (Active Comparator): To prevent agitation deksmedetomidine infused during operation and at the end of surgery agitation scor measured by Riker sedation agitation scale.
  Interventions: Drug: deksmedetomidine
- Remifentanil infusion (Experimental): To prevent agitation remifentanil infused during operation at the end of surgery agitation scor measured by Riker sedation agitation scale.
  Interventions: Drug: Remifentanil
- Saline infusion (Placebo Comparator): Saline infused during operation and at the end of surgery agitation scor measured by Riker sedation agitation scale.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: deksmedetomidine — deksmedetomidine infused during operation 0.2 mcg/kg/hour
  Other Names: Precedex
  Arms: Deksmedetomidine infusion
Drug: Remifentanil — Remifentanil infused during operation 0.2 mcg/kg/min
  Other Names: Ultiva
  Arms: Remifentanil infusion
Drug: Saline — During operation saline infused equal volüme of deksmedetomidine and remifentanil
  Arms: Saline infusion

SUMMARY:
To compare the effect of two different agents deksmedetomidine, remifentanil and placebo, agitation and recovery condition, on nasal septum operation.

DETAILED DESCRIPTION:
Nasal septum operation cause agitation because of nasal package. This research aims determine which agent , deksmedetomidine remifentanil or placebo, is more beneficial to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients

Exclusion Criteria:

* patients with any sensitivity each drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To asses postoperative agitation score by Riker sedation agitation scale | Postoperative first hour

SECONDARY OUTCOMES:
Yo asses postoperative side effects emesis, vomitting or pain | Postoperative first hour

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Polat, MD, Principal Investigator — Yildirim Beyazit Education and Research Hospita
Locations (1):
- Reyhan Polat, Ankara, Turkey (Türkiye)